CLINICAL TRIAL: NCT05658471
Title: Comparative Pharmacokinetics and Pharmacodynamics of Nicotine With Use of NIDA Standardized Research Electronic Cigarette (SREC) vs Usual Brand E-cigarette
Brief Title: Pharmacokinetics and Pharmacodynamics of Nicotine With Use of Standardized Research Electronic Cigarette (SREC)
Acronym: SREC22
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SREC22; 5U01DA045519-02 (NIH)
Record Dates: First submitted 2022-12-09; First posted 2022-12-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Nicotine Dependence; Tobacco Toxicity; Cardiovascular Risk Factors
Keywords: Nicotine Pharmacokinetics; Nicotine Pharmacodynamics; Electronic Cigarettes; E-Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the starting condition using a Latin square design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Brand E-Cigarette (EC) then SREC (Experimental): Participants will be admitted to hospital research ward within 32 hours of the orientation visit and begin a standardized session of product use using the usual brand of e-cigarette that participants utilize for nicotine use, and will provide expired carbon dioxide samples, pharmacokinetic (PK) blood samples, urine samples, and have cardiovascular and vital signs monitored. Participants will also be asked to complete nicotine-related questionnaires. Participants will then return within 2 weeks to repeat the procedures using the SREC.
  Interventions: Other: Standardized Research E-Cigarette (SREC); Other: Over the Counter E-Cigarette (EC); Behavioral: Biological Samples; Other: Smoking-related Questionnaires
- SREC then Usual Brand E-Cigarette (EC) (Experimental): Participants will be admitted to hospital research ward within 32 hours of the orientation visit and begin a standardized session of product use using the SREC, and will provide expired carbon dioxide samples, pharmacokinetic (PK) blood samples, urine samples, and have cardiovascular and vital signs monitored. Participants will also be asked to complete nicotine-related questionnaires. Participants will then return within 2 weeks to repeat the procedures using the usual brand of e-cigarette that participants utilize for nicotine use.
  Interventions: Other: Standardized Research E-Cigarette (SREC); Other: Over the Counter E-Cigarette (EC); Behavioral: Biological Samples; Other: Smoking-related Questionnaires

INTERVENTIONS:
Other: Standardized Research E-Cigarette (SREC) — Standardized Research E-Cigarette (SREC) will be obtained through NJOY, LLC and provided at the hospital stay.
Other: Over the Counter E-Cigarette (EC) — Usual brand e-cigarettes will be provided at the hospital stay.
  Other Names: Usual Brand E-Cigarette (EC)
Behavioral: Biological Samples — Blood, urine, and expired carbon dioxide will be obtained during the course of the study.
  Other Names: Biological Specimens
Other: Smoking-related Questionnaires — Nicotine and Smoking behavior and dependence questionnaires will be administered at screening, before and during hospital stays.
  Other Names: Behavioral Questionnaires

SUMMARY:
This is a crossover study that will examine use behaviors, chemical exposures, and biological effects of Standardized Research Electronic Cigarette (SREC) compared to usual brand e-cigarette use in natural or synthetic nicotine users.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To characterize nicotine delivery, systemic exposure and effects from SREC in comparison with usual to usual nicotine brand use.

II. To assess aspects of harm of SREC use compared to usual nicotine brand use.

OUTLINE:

Eligible participants will be assigned to one of two treatment conditions for the initial assessment which will take place in a hospital setting. The participant will then be assigned to the second condition within 2 weeks after the initial assessment which will also take place in a hospital setting to repeat the same procedures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history and limited physical examination-

  * Heart rate < 105 beats per minute (BPM)*.
  * Systolic Blood Pressure < 160 and > 90*.
  * Diastolic Blood Pressure < 100 and > 50*.
  * *considered out of range if both machine and manual readings are above/below these thresholds.
  * Body Mass Index <= 38.0.
* Current regular user of electronic cigarettes (EC)

  * EC device use at least 15 or more days in the past 30 days (with e- liquid >= 3mg/ml)
  * No restriction on flavor or type of e-cigarette used
  * Saliva cotinine >= 50 ng/ml and/or NicAlert = 6
* Age >= 21 years old <= 70 years old
* Willingness to abstain from drug use for the duration of the study

Exclusion Criteria:

* The following unstable medical conditions:

  * Heart disease
  * Seizures
  * Cancer
  * Thyroid disease (okay if controlled with medication)
  * Diabetes
  * Hepatitis B or C or Liver disease
  * Glaucoma
  * Kidney disease or urinary retention
  * History of stroke
  * An ulcer in the past year
  * Active use of an inhaler for Asthma or chronic obstructive pulmonary disease (COPD)
* Medications

  * Use of medications that are inducers of nicotine metabolizing enzyme CYP2A6 (Example: rifampicin, carbamazepine, phenobarbital, and other anticonvulsant drugs).
  * Use of sympatholytic medications for cardiovascular conditions including hypertension (Example: beta and alpha-blockers).
  * Concurrent use of nicotine-containing medications (Example: nicotine patch, lozenge, gum).
  * Any stimulant medications (example: Adderall) generally given for attention deficit hyperactivity disorder (ADHD) treatment.
* Other/Misc. Health Conditions

  * Oral thrush
  * Fainting (within the last 30 days)
  * Other "life threatening illnesses" as per principal investigator and/or study physician's discretion
* Pregnancy

  * Pregnancy (self-reported and urine pregnancy test)
  * Breastfeeding (determined by self-report)
  * Women of childbearing potential must be using an acceptable method of contraception
* Concurrent participation in another clinical trial.
* Inability to read and write in English
* Planning to quit smoking or vaping within the next 60 days
* A known propylene glycol/vegetable glycerin allergy
* Uncomfortable with getting blood drawn
* Recent onset or change (worsening) in cough, fever and/or abdominal symptoms (vomiting or pain) in the past two weeks

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean Peak Nicotine Concentration | Collected 2, 5, 7, 10, 15, 30, 45, 60, 75, 90, and 120 minutes post end vaping session
  The investigators will compare peak nicotine concentrations between SREC vs. EC use
Mean Time of Peak Nicotine Concentration | Collected 2, 5, 7, 10, 15, 30, 45, 60, 75, 90, and 120 minutes post end vaping session
  Compare peak nicotine concentration between SREC vs. EC use.
Area Under the plasma nicotine concentration-time Curve (AUC) at 120 minutes | Collected 2, 5, 7, 10, 15, 30, 45, 60, 75, 90, and 120 minutes post end vaping session
  Compare peak nicotine concentration between SREC vs. EC
Mean overall systemic nicotine exposure | during the 3 hr of ad libitum use
  Descriptive statistics will be used to examine systemic nicotine exposure from use of SREC and compare to EC
Mean inter-puff interval | during the 3 hr of ad libitum use
  The patterns of SREC puffing and EC use will be examined looking at the average and variability (SD) of inter-puff interval during the 3 hr of ad libitum use.
Change in Mean score on the Modified Cigarette Evaluation Questionnaire (mCEQ) | Up to 1 month
  The mCEQ use three multi-item domains (subscales) and two single items: "Smoking Satisfaction", "Psychological Reward", "Aversion", "Enjoyment of Respiratory Tract Sensations" and "Craving Reduction". Scores for each subscale are calculated as the average of its individual item responses of The items are rated on a seven-point scale ranging from 1 (not at all) to 7 (extremely). Higher scores indicate greater intensity of each smoking effect with, for example, greater satisfaction or psychological reward after smoking. Scores will be compared between SREC and EC use.
Change in Mean score on the Minnesota Tobacco Withdrawal Scale-Revised (MTWS-R) | Up to 1 month
  The MTWS-R features two separate measures for examining the severity of nicotine withdrawal symptoms in a participant: a self-report scale and an observer scale. The observer scale asks the scale-taker to rate the severity of four symptoms in someone the they know who is experiencing nicotine withdrawal: "angry/irritable/frustrated," "anxious/tense," "depressed," and "restless/impatient." The self-report version asks for rankings of the severity of those same four symptoms, plus eleven others that cannot be observed by outsiders (including such things as "desire or craving to smoke," "insomnia, sleep problems, awakening at night," or "dizziness). Both scales use a Likert-type scale for the severity ratings, ranging from 0 ("not at all") to 4 ("severe"). These scores are tallied to calculate an a total withdrawal discomfort score and will be compared between SREC and EC use
Change in Mean score on the Questionnaire on Smoking Urges (QSU-Brief) | Up to 1 month
  The QSU-Brief consists of 10 statements about the respondent's feelings and thoughts about the participants desire to smoke cigarettes as the participant is completing the questionnaire (i.e., right now). Each response is scored a number ranging from 1 (strongly disagree) to 7 (strongly agree) and total scores are calculated by summing the item scores to compare craving between SREC and EC use

SECONDARY OUTCOMES:
Mean acrolein levels within participants | Up to 1 month
  Urine excretion of mercapturic acid metabolites of volatile organic compounds (VOCs), with a particular focus on acrolein will be measured and compared between SREC and EC use
Mean propylene oxide levels within participants | Up to 1 month
  Urine excretion of mercapturic acid metabolites of VOCs, with a particular focus on propylene oxide will be measured and compared between SREC and EC use
Median benzene levels within participants | Up to 1 month
  Urine excretion of mercapturic acid metabolites of VOCs, with a particular focus on benzene will be measured and compared between SREC and EC use
Mean heart rate within participants | Up to 1 month
  The cardiovascular effects of e-cigarette use as measured by heart rate will be compared between SREC and EC use
Mean blood pressure (both systolic and diastolic) within participants | Up to 1 month
  The cardiovascular effects of e-cigarette use as measured by blood pressure will be compared between SREC and EC use
Mean plasma epinephrine within participants | Up to 1 month
  The cardiovascular effects of e-cigarette use as measured by plasma epinephrine will be compared between SREC and EC use

CONTACTS AND LOCATIONS:
Overall Officials: Neal Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco - Tobacco Research Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No